CLINICAL TRIAL: NCT04255823
Title: Efficacy of a Multi-faceted Intervention to Deprescribe Proton Pump Inhibitors (PPI) in Primary Care: a Population-based, Pragmatic, Cluster-randomized Controlled Trial.
Acronym: DeprescrIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RC19_0460
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Proton Pump Inhibitors; Deprescription
Keywords: Proton pump inhibitors; Deprescription; Multi-faceted intervention; Patient-centered; Primary health care; Pharmacoepidemiology
MeSH Terms: interventions — General Practitioners

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multi-faceted intervention (Experimental): A patient education material on PPI deprescribing will be send to patients with long-term treatment with PPI (>300DDD/patient/year).
  Their general practitioner (GP) will receive a "dear doctor" letter with an algorithm related to PPI deprescribing.
  Interventions: Other: General practitioner and Patient receive informations related to PPI deprescribing.
- "Dear doctor" letter of the GP (Experimental): Only the GP will receive the "dear doctor" letter with the algorithm.
  Their patients will not receive any patient education material.
  Interventions: Other: Only General practitioner receive informations related to PPI deprescribing.
- Control (No Intervention): Neither the patients nor their GP will receive information.

INTERVENTIONS:
Other: General practitioner and Patient receive informations related to PPI deprescribing. — General practitioner will receive a sensibilization and an algorithm related to PPI deprescribing.
  Their patients will receive any informations (patient information material on PPI deprescribing)
  Arms: Multi-faceted intervention
Other: Only General practitioner receive informations related to PPI deprescribing. — General practitioner will receive the sensibilization and an algorithm related to PPI deprescribing.
  Their patients will not receive any informations.
  Arms: "Dear doctor" letter of the GP

SUMMARY:
Deprescribing is defined as "the process of withdrawal of an inappropriate medication, supervised by a health care professional with the goal of managing the polypharmacy and improving outcomes". Inappropriate use of proton pump inhibitors (PPI) is associated with severe adverse drug reactions and a major economic impact. Deprescribing should be considered when inappropriate prescription of PPI is identified.

DeprescrIPP is a pragmatic population-based cluster-randomized trial conducted in primary care. It will assess the efficacy and effectiveness of a multi-faceted intervention (on patients and general practitioners) to deprescribe PPI.

ELIGIBILITY:
Inclusion Criteria:

* General practitioners (GPs):

  • All GPs settled in the 2 departments of Loire-Atlantique and Vendée with more than 100 patients in the year before baseline, will be eligible.
* Patients:

  * aged over 18 years
  * affiliated to the French health insurance system (CPAM)
  * treated with PPI with more than 300 DDD/year in the year before baseline, estimated with reimbursement databases.
  * whose GP is included in the study

Exclusion Criteria:

* General practitioners (GPs):

  • Participation refusal
* Patients :

  * Participation refusal
  * Patients at risk of gastroduodenal lesions i.e. treated with nonsteroidal anti-inflammatory drugs (NSAIDs) and over 65 years old or treated with either corticosteroids or anticoagulants or platelet aggregation inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34000 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
PPI deprescribing | 12 months
  Proportion of patients achieving a 50% decrease in their reimbursement of PPI (Defined Daily Dose (DDD)/year) at the end of the intervention compared to baseline.

SECONDARY OUTCOMES:
Cost-utility analysis | 12 months
  Incremental cost-utility ratio (cost by quality-adjusted life-years, QALY) of control group compared to the intervention.
GERD symptoms recurrence | 12 months
  A short-form REFLUX-QUAL questionnaire will be assessed to a 10% patient sample in each arm (baseline and 12 months)
Attitudes of patients towards deprescribing | 12 months
  Revised patients' attitudes toward deprescribing questionnaire will be assigned to a 10% patient sample in each arm (baseline and 12 months)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen-Soenen J, Rat C, Gaultier A, Schirr-Bonnans S, Tessier P, Fournier JP. Effectiveness of a multi-faceted intervention to deprescribe proton pump inhibitors in primary care: protocol for a population-based, pragmatic, cluster-randomized controlled trial. BMC Health Serv Res. 2022 Feb 17;22(1):219. doi: 10.1186/s12913-022-07496-3. PMID 35177042